CLINICAL TRIAL: NCT04103840
Title: Assessment of Invasive Fungal Infections as a Result of Fungal Dysbiosis in Patients With Severe Alcohol-associated Hepatitis
Brief Title: Invasive Fungal Infections in Severe Alcohol-associated Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC-08/2019-1270
Record Dates: First submitted 2019-09-01; First posted 2019-09-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Severe Alcoholic Hepatitis; Chronic Liver Disease and Cirrhosis
MeSH Terms: conditions — Hepatitis, Alcoholic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal mycobiota
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe alcohol- associated hepatitis: Severe alcohol associated hepatitis as defined by probable/ conformed National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria
  Interventions: Other: Testing stool mycobiota
- Control: Apparently healthy Family controls
  Interventions: Other: Testing stool mycobiota

INTERVENTIONS:
Other: Testing stool mycobiota — Both cohorts of SAH and their family controls will be tested for fecal mycobiota

SUMMARY:
Chronic alcohol consumption is associated with intestinal bacterial dysbiosis, yet little is known about the role of intestinal fungi, or mycobiota in liver disease. Although the intestinal microbiome contains bacteria, fungi, and viruses, research in the field of liver disease has almost exclusively focused on the interaction between the host and gut bacteria. The fungal microbiota is an integral part of the gastrointestinal micro-ecosystem with up to 106 microorganisms per gram of faeces. Numerous interactions between fungi and bacteria and the complex immune response to gastrointestinal commensal or pathogenic fungi have been demonstrated in prior studies. Alcohol-dependent patients display a reduced intestinal fungal diversity and Candida overgrowth. Compared with healthy individuals and patients with non-alcohol-related cirrhosis, alcoholic cirrhosis patients also demonstrate systemic exposure and immune response to mycobiota. Thus, chronic alcohol consumption is associated with an altered mycobiota and translocation of fungal products. Manipulating the intestinal mycobiome might be an effective strategy for attenuating alcohol-related liver disease especially alcoholic hepatitis. In this study, we will attempt to find out the natural fungal mycobiome in Severe alcoholic hepatitis when compared with apparently healthy asymptomatic controls from their family. This will allow us to therapeutically modify the unbalanced gut microbiota and improve patient outcomes. Secondly, it will provide further insight as to why alcohol-associated hepatitis patients are particularly susceptible to fungal infections. In the age of frequent antibacterial drug therapy, the role of commensal and pathogenic fungi in the human gut has gained paramount importance.

DETAILED DESCRIPTION:
The patients of severe alcohol-associated hepatitis admitted under Department of Hepatology, in Liver intensive Care Unit (LICU) Male or Female medical wards or coming to follow up in Liver clinic of Postgraduate Institute of Medical Education and Research, Chandigarh, India from will be screened for enrolment after ethical approval from the institute ethics committee. Both previously compensated and decompensated patients will be enrolled in this prospective observational pilot study. All patients will be followed up at 30 and 90 days from inclusion into the study.

Estimation of sample size Sample size will be estimated based on previous studies. This is a pilot prospective observational study. Based on currently available data from our centre on acute-on chronic liver failure, 22.5% of cirrhotics have suspected IFI, and up to 25% of SAH have suspicion for IFI, it is estimated that a total sample size of 60 patients would be required, with an effect size of 0.5, alpha 0.05, and power 0.85. Therefore, 80 patients will be required to enroll to account for 15% attrition. Hence, we propose to enroll 80 consecutive patients with SAH with 80 matched controls from their family starting from 15th August 2019.

ELIGIBILITY:
Inclusion Criteria:

* Severe Alcoholic Hepatitis
* Aged between 18 Years to 70 Years
* Either gender
* Study will also include age matched healthy controls from the patient's family

Exclusion Criteria:

1. Inability to obtain informed consent from patient or relatives.
2. Severe cardiopulmonary disease
3. Pregnancy
4. HIV infection
5. Recent abdominal surgery (with in last 6 months)
6. Patient on immunosuppressive drugs
7. Malignancies including Hepatocellular carcinoma
8. Gastrointestinal (GI bleed) in the last 4 weeks
9. Oral antibiotics or antifungals taken in last 2 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alcohol-associated hepatitis (AH) is defined by National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria as biopsy proven or clinically diagnosed AH in patients with heavy alcohol use and typical liver tests without confounding factors
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | at Day 28 and Day 90
  Patients who survive till Day 28 and Day 90

SECONDARY OUTCOMES:
Non-elective hospital admissions | 90 Days
  Number of hospital admissions will be documented
Clinical and biochemical parameters will be compared at 0 and 90 days | 90 days
  Change in biochemical parameters including liver function tests, renal function tests, ammonia etc.
Clinical events like decompensation in the form of new onset ascites, variceal bleed, renal dysfunction, hepatic encephalopathy, infections | 90 days
  Number of decompensation events [ascites, variceal bleed, renal dysfunction, hepatic encephalopathy, infections]

CONTACTS AND LOCATIONS:
Overall Officials: Radha Dhiman, MD DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided